CLINICAL TRIAL: NCT03302338
Title: Simulated Amniotic Fluid Like Solution Enterally Administrated in Neonates Recovering From GIT Surgeries
Brief Title: Simulated Amniotic Fluid Solution in Neonates Recovering From GIT Surgeries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rania Ali El-Farrash (Other)
Responsible Party: Sponsor-Investigator, Rania Ali El-Farrash, Clinical Professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SAFE 2013
Record Dates: First submitted 2015-05-17; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Necrotizing Enterocolitis
Keywords: Feeding intolerance; Simulated amniotic fluid like solution; Necrotizing enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAFE group (Experimental): SAFE group: simulated amniotic fluid 20cc/kg/day enterally divided according to number of feds (syringe for every fed). This amount provides enteral 4.5μg rhG-CSF / kg/day and enteral 88IU rhEPO / kg/day.
  Interventions: Drug: SAFE group
- Placebo (Placebo Comparator): Placebo group: distilled water 2.5 ml/kg every 3 hours enterally given.
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: SAFE group — simulated amniotic fluid 20cc/kg/day enterally for a maximum of 7 days.
  Other Names: simulated amniotic fluid like solution 20cc/kg/day enterally
  Arms: SAFE group
Drug: placebo group — distilled water 20 ml/kg/day for maximum of 7 days.
  Other Names: distilled water
  Arms: Placebo

SUMMARY:
Amniotic fluid plays a significant role in fetal gut maturation and development. The human fetus swallows over 200 ml of amniotic fluid per kilogram of weight each day and such swallowing is essential for normal small bowel development.Growth factors found in the amniotic fluid have been shown to promote proliferation of fetal intestinal cells. As feeding intolerance is a common problem among neonates recovering from surgery for congenital bowel abnormalities, the investigators will study the role of enteral administration of simulated amniotic fluid solution in prevention of feeding intolerance and NEC in neonates recovering from GIT surgeries.

DETAILED DESCRIPTION:
Neonates with congenital GIT anomalies will participate after being operated.

Participants will be followed for the duration of hospital stay until discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with operable congenital bowel abnormalities

Exclusion Criteria:

* Critically ill babies.
* Presence of any contraindications to enteral feeding

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Signs of feeding intolerance | through study completion, an average of 1 year
  Feeding intolerance defined as distended loops of bowel, bilious vomiting, large pre-feeding gastric residuals more than 20% of each feed, diarrhea, occult or gross blood in stools, abdominal wall erythema or ecchymosis

SECONDARY OUTCOMES:
Necrotizing enterocolitis | The outcome measure will be assessed within 2 months
  • Clinical signs of suspected NEC (abdominal distension, increased volume of gastric aspirate, bile stained aspirate, and / or apnea or bradycardia), and Bell's modified criteria for staging (Bell et al., 1978).
hospital stay | through study completion, an average of 1 year
  duration on hospitalization
mortality | he outcome measure will be assessed within 2 months
  death

CONTACTS AND LOCATIONS:
Overall Officials: Rania A El-Farrash, MD, Study Director — ASU
Locations (1):
- Ain Shams University, Cairo, Egypt